CLINICAL TRIAL: NCT04310475
Title: Virtual Reality Assisted CBT for Social Difficulties: a Feasibility Study in Early Intervention for Psychosis Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Lucia Valmaggia, Reader in Clinical Psychology and Digital Mental Health, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 255964
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Psychosis; Social Behavior; Paranoia; Social Anxiety
MeSH Terms: conditions — Psychotic Disorders; Social Behavior; Paranoid Disorders

STUDY DESIGN:
Intervention Model Description: Case series, feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental): This is a case series
  Interventions: Other: Virtual reality assisted CBT

INTERVENTIONS:
Other: Virtual reality assisted CBT — This study uses virtual reality technology to assist cognitive behavioural therapy for social difficulties in people with first episode psychosis.

SUMMARY:
People experiencing psychosis might find social interactions stressful and avoid them. This can result in isolation and can affect relationships, employment and quality of life. Improving social functioning is a really important aspect of recovery. Facing social situations after the first episode of psychosis can be very difficult and provoke intense anxiety. However, research has shown that the earlier intervention is offered, the better the outcome. Therefore, improving therapies for people experiencing their first episode of psychosis is a key target for research. Virtual Reality presents a unique opportunity to bring real-life-type environments into a therapy session to help people to overcome their distress in social situations and make them feel less anxious. Virtual Reality assisted Therapy (VRT) provides a 'safe space' to practice strategies and techniques to help people work towards improving their social functioning, build new ways of coping with stress and assist them in their recovery.

The study uses a standard CBT model and integrates a Virtual Reality environment into it to support exposure and behavioural experiments for social difficulties, which are a key component of treatment.

DETAILED DESCRIPTION:
Participants will be offered up to 10 sessions including a pre and post assessment session. Each participant will set one or more SMART goals for therapy (e.g. be able to use public transport, attend a social gathering or to feel less anxious in social situations) which are worked on both in the therapy sessions and through homework tasks.

This is a feasibility study. The aim is to recruit between 6-10 participants to pilot the VRT with. The results of this study will inform future research and practice, by helping to assess if service-users find the new VRT acceptable (e.g. recruitment, retention, drop out rates, participant experiences), and if it is effective (e.g. reduction in symptoms or distress, and improvement in social functioning).

It is really important that the clinical care of anyone who chooses to participate in the study is not affected by their participation in this study. The researchers will work closely with clinical teams to ensure this. Clients who engage with the study will still be eligible for all aspects of TAU including psychological interventions, should this be appropriate.

The VR technology and environment has been used extensively before in research studies, which have proved that it is safe and effective. However, it has not been used within the NHS context before or embedded within a therapy course before.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be under the care of an approved research site throughout the period of the study i.e. local early intervention for psychosis clinical team
* The participant must be aged 18-65 and speak English to a conversational level.
* The participant must have experienced or currently be experiencing psychosis, as defined by ICD-10 and DSM-V criteria.
* The participant must have the capacity to consent to the study
* The participant should be experiencing difficulties in social situations (e.g. due to paranoia, social anxiety, poor social skills, low mood or lack of social motivation)

Exclusion Criteria:

* The participant must not have a history of epilepsy OR photosensitivity (any other comorbidity is fine).
* The participant must not currently be in receipt of another psychological therapy at the time of the study (before or after the study is fine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention | From start of study until completion of recruitment, approximately 8 months
  To assess feasibility and acceptability data will be collected regarding the number of people approached, engaged, dropped out, completed the intervention
Qualitative feedback from clients and therapists about their experiences | From start of study until completion of intervention, approximately 10 months
  To assess feasibility and acceptability feedback from clients and therapists about the experience of the receiving and/or delivering the intervention will be regularly sought via interview.
Study resources | From start of study until completion of intervention, approximately 10 months
  To assess feasibility and acceptability the resources required for the intervention will be recorded (e.g. from training and supervising therapists, to room space, technological kit and support required etc.) as observations.

SECONDARY OUTCOMES:
Pre and post therapy psychometric assessment - mood | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in mood before and after receiving the intervention using the PHQ-8 (a self report questionnaire measure of depression).
Pre and post therapy psychometric assessment - anxiety | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in anxiety before and after receiving the intervention using the GAD-7 (a self report questionnaire measure of generalised anxiety).
Pre and post therapy psychometric assessment - social anxiety 1 | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in social anxiety before and after receiving the intervention using the Social Anxiety and Distress Scale (SADS; a self report questionnaire measure of social anxiety and distress).
Pre and post therapy psychometric assessment - social anxiety 2 | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in social anxiety before and after receiving the intervention using the Brief Fear of Negative Evaluation (BFNE; a self report questionnaire measure of fear of negative evaluation in the context of social anxiety).
Pre and post therapy psychometric assessment - paranoid thoughts | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in paranoid thoughts before and after receiving the intervention using the Green Paranoid Thoughts Scale (GPTS; a self report questionnaire measure of paranoid thoughts).
Pre and post therapy psychometric assessment - interpersonal sensitivity | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in interpersonal sensitivity before and after receiving the intervention using the Interpersonal Sensitivity Measure (IPSM; a self report questionnaire measure of interpersonal sensitivity).
Pre and post therapy psychometric assessment - symptom related distress | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in symptom related distress before and after receiving the intervention using the CORE-10 (a self report questionnaire measure of symptom related distress).
Pre and post therapy psychometric assessment - loneliness | Start and end of each individual intervention at approximately 10-16 week interval, up to 10 months
  To assess the potential intervention efficacy, psychometric data will be collected pre and post intervention to assess change in experience of loneliness before and after receiving the intervention using the UCLA Loneliness scale (UCLAL-20; a self report questionnaire measure of interpersonal sensitivity).
Progress towards individualized SMART goal | Start, middle and end of each individual intervention within approximately 10-16 week window, up to 10 months
  To assess the potential intervention efficacy, clients will set a SMART goal to work on during therapy. Progress towards achieving this goal will be assessed using scaling questions throughout therapy.
Adverse effects | At completion of each intervention or when clients drop out from the study, up to 10 months
  To assess for any potential adverse effects of the intervention, e.g. increase in symptoms/ reduction in functioning, clients will be asked to complete a questionnaire assessing this at the end of the intervention or if they drop out from the study. This questionnaire has been co-developed with a peer researcher for the purposes of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No